CLINICAL TRIAL: NCT03467711
Title: The Use of Tidal Volume Challenge to Improve the Reliability of Dynamic Parameters (Pulse Pressure Variation and Stroke Volume Variation) During Pneumoperitoneum and Laparoscopic Surgery
Brief Title: The Use of Tidal Volume Challenge of Dynamic Parameters During Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, Assistant Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: 2017-009-003-002
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tidal volume challenge — transiently increasing tidal volume from 6 to 8 mL/kg predicted body weight (tidal volume challenge)
Other: volume expansion — give 6ml/kg (predicted body weight) volulyte for 10min

SUMMARY:
Laparoscopy is increasingly used for major abdominal and pelvic surgery. As this approach is also recommended in elderly patients with serious comorbidities, optimal fluid therapy guidance during this procedure is important.

Many studies have reported that less invasive dynamic indices such as pulse pressure variation (PPV) and stroke volume variation (SVV), which are derived from the arterial pressure waveform, are superior to static indices to predict fluid responsiveness. PPV and SVV are based on the heart-lung interaction and reflect cyclic changes in stroke volume induced by mechanical ventilation in the closed-chest condition. Therefore, their ability to predict fluid responsiveness can be affected by factors that influence the arterial tone or the compliance of the respiratory system.

Laparoscopic surgery for the abdominal visceral organs requires pneumoperitoneum and the Trendelenburg position to optimize surgical conditions, and can reduce cardiac output and respiratory compliance. Accordingly, the usefulness of PPV and SVV in predicting fluid responsiveness during laparoscopic surgery under these conditions may be questioned.

It has been clearly shown that the values of dynamic parameters are significantly correlated with the magnitude of VT. Min et al. reported that augmentation of PPV and SVV via a temporary increase in VT from 8 to 12 ml/kg improved their predictive power in the inconclusive zone with respect to fluid responsiveness (PPV values of 9% and 13%, respectively). Another recent study reported that on increasing VT from 6 to 8 ml/kg, augmented PPV and SVV, as well as their absolute changes, predicted fluid responsiveness with high sensitivity and specificity, even in critically ill patients receiving low VT.

Therefore, the aim of the current study was to investigate whether increasing VT from 6 to 8 ml/kg would improve the predictive power of PPV and SVV in patients undergoing robot-assisted laparoscopic surgery in the Trendelenburg position under lung-protective ventilation. We also assessed the ability of absolute changes in PPV and SVV values induced by a temporary increase in VT from 6 to 8 ml/kg to predict fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who performed robot assisted laparoscopic surgery under Trendelenburg position

Exclusion Criteria:

* preoperative arrhythmia
* Severe bradycardia
* Moderate to severe valvular disease
* left ventricular ejection fraction < 50%
* Poorly controlled hypertension (systolic BP > 160 mmHg)
* Patients with renal insufficiency (creatinine > 1.5 mg/dL)
* Moderate to severe liver disease
* BMI >.30 or < 15 kg/ m2
* preexisting pulmonary disease
* FEV1 < 60% of predicted value
* contraindications to oesophageal Doppler (OED) monitoring probe insertion (i.e. oesophageal stent, carcinoma of the oesophagus or pharynx, previous oesophageal surgery, oesophageal stricture, oesophageal varices, pharyngeal pouch, and severe coagulopathy)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary care center
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
PPV8 | 3min after tidal volume challenge
  augmented pulse pressure variation using a temporary increase in VT
SVV8 | 3min after tidal volume challenge
  augmented stroke volume variation using a temporary increase in VT

SECONDARY OUTCOMES:
ΔPPV6-8 | 3min after tidal volume challenge
  The changes in pulse pressure variation obtained by transiently increasing tidal volume
ΔSVV6-8 | 3min after tidal volume challenge
  The changes in stroke volume variation obtained by transiently increasing tidal volume
PPV6 | Before fluid expansion
  The value of pulse pressure variation when protective ventilation applied
SVV6 | Before fluid expansion
  The value of stroke volume variation when protective ventilation applied
PPV_fb | 5min after fluid expansion
  The change in PPV after giving the fluid expansion
SVV_fb | 5min after fluid expansion
  The change in SVV after giving the fluid bolus

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jun JH, Chung RK, Baik HJ, Chung MH, Hyeon JS, Lee YG, Park SH. The tidal volume challenge improves the reliability of dynamic preload indices during robot-assisted laparoscopic surgery in the Trendelenburg position with lung-protective ventilation. BMC Anesthesiol. 2019 Aug 7;19(1):142. doi: 10.1186/s12871-019-0807-6. PMID 31390982